CLINICAL TRIAL: NCT00271700
Title: Improving Glycemic Control on GMS: A Quality Improvement Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Jeffrey Schnipper, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-P-001880/1; 2005-P-001880/1
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Outcome Assessment (Healthcare); Inpatients; Hospital Information Systems; Education
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Usual Care (No Intervention): admission to medical team floor to usual care
- Intervention (Experimental): consists of usual care as well as an admission order set built into BWH's proprietary computer provider order entry (CPOE) system
  Interventions: Behavioral: Order Set, Education, Feedback

INTERVENTIONS:
Behavioral: Order Set, Education, Feedback
  Arms: Intervention

SUMMARY:
This study will examine whether new processes and technologies for monitoring diabetic patients' insulin levels improves patient care at Brigham and Women's Hospital.

DETAILED DESCRIPTION:
This study will examine whether new processed and technologies for monitoring diabetic patients' insulin levels improves patient care. Patients at Brigham and Women's Hospital (BWH), staying on the General Medicine Service, who have Type 2 diabetes and who are not on IV insulin can participate in this study. Physicians and nurses will be taught new rules to care for diabetic patients, while in the hospital. Also, the BWH computer system will be updated to include these new rules for administering insulin. Patients who participate in the study will be randomly placed into one of two groups: one group that will be cared for by physicians and nurses who have learned these new rules for administering insulin; or the second group, who will receive diabetes care at BWH before the new rules were adopted. The study will last approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include all type 2 diabetic patients on the General Medicine Service (GMS) of Brigham and Women's Hospital (BWH) who do not have an indication for IV insulin.

Exclusion Criteria:

* Type 2 diabetic patients on the General Medicine Service (GMS) of Brigham and Women's Hospital (BWH) who have an indication for IV insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
- Point-of-care testing glucose values (percent of routine glucose readings between 60 and 180 mg/dL)
- Lab glucose values (percent of routine glucose readings between 60 and 180 mg/dL)

SECONDARY OUTCOMES:
- Quality of insulin orders using explicit criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States